CLINICAL TRIAL: NCT00009594
Title: Alternative Medicine Approaches for Women With Temporomandibular Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Purpose: Diagnostic
Other Study IDs: P50AT000076-01P2 (NIH); P50AT000076-01 (NIH); NCT00009282 (obsolete NCT alias)
Record Dates: First submitted 2001-02-01; First posted 2001-02-02 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Naturopathy; Medicine, Chinese Traditional

INTERVENTIONS:
Procedure: Naturopathic Medicine
Procedure: Traditional Chinese Medicine

SUMMARY:
Temporomandibular disorders (TMD) are characterized by pain and tenderness in the muscles of mastication and/or the temporomandibular joint (TMJ), limitations of jaw opening often accompanied by deviations in mandibular path, and clicking, popping or grating TMJ sounds.

TMD is often found in association with other problems: depression, anxiety, sleep disturbances, gastrointestinal symptoms, frequent infections, etc. This project proposes to holistically address patient symptoms through three different approaches, Naturopathic Medicine (NM), Traditional Chinese Medicine (TCM), and usual care at KPNW. We will conduct a pilot test and Phase II trial to evaluate the two alternative healing approaches, TCM (n=50) and NM (n=50) delivered by TCM and NM practitioners, are as effective as usual TMD care (n=50) provided by dental clinicians in the KPNW TMD Clinic. Subjects will be females 25-55 years of age with multiple health problems (defined as patients who have had at least 4 organ system-grouped diagnoses in the past year, not including TMD). Subjects will be evaluated at baseline, 6 and 12 months after start of treatment. The primary endpoint is change from baseline in the Axis II Pain Related Disability and Psychological Status Scale. Clinical examinations, saliva samples to assess salivary cortisol levels, and responses to a series of questionnaires to assess pain, chronic pain, psychosocial functioning, and other physical symptoms will be used to assess outcomes. We will passively monitor health care utilization within KPNW using clinical, research, and administrative databases to determine whether the interventions have an impact on overall health care utilization. If either of these alternative interventions is shown to merit Phase III trial, our goal is to design and implement such a clinical trial to further evaluate the health consequences and costs of these alternative healing paradigms.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
- Patients who have had at least 4 organ system-grouped diagnoses in the past year, not including TMD

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-09; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Alexander White, Principal Investigator — Center for Health Research (CHR), Kaiser Foundation Hospitals
Locations (1):
- Center for Health Research, Kaiser Foundation Hospitals, Portland, Oregon, United States